CLINICAL TRIAL: NCT07156838
Title: Evaluation of Bioflex and Zirconia Crowns Versus Stainless Steel Crowns on Primary Molars: Randomized Controlled Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Asmaa Yahia, BDS, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1003-11/2024
Record Dates: First submitted 2025-08-27; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Badly Decayed Primary Molars; Preformed Pediatric Posterior Crowns
Keywords: bioflex crown; zerconia crown; stainless steel crown; clinical success

STUDY DESIGN:
Masking Description: Data analyst
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- bioflex crown (Experimental)
  Interventions: Other: bioflex crown
- zerconia crown (Experimental)
  Interventions: Other: zerconia crown
- stainless steel crown (Active Comparator)
  Interventions: Other: stainless steel crown

INTERVENTIONS:
Other: bioflex crown — A preformed bioflex crown of similar size will be selected. Tooth preparation will be done using a tapered diamond bur to reduce the occlusal surface, including the central groove, by 1-1.5 mm. The proximal surfaces will be prepared by approximately 0.5 mm to clear the contact area, bioflex crown fitting and proper occlusion will be checked then it will be cemented using type-I glass ionomer cement, Any excess cement will be removed.
  Arms: bioflex crown
Other: zerconia crown — Occlusal reduction will be done by 1-1.5 mm using coarse football shaped diamond bur following the natural occlusal anatomy.
  Interproximal contacts will be opened with a tapered fissure bur. The proximal space should be enough to permit the chosen crown to fit passively.
  The molar will be trimmed down circumferentially 0.5-1.25 mm as needed with the use of tapered diamond burs.
  •About 1 to 2 mm subgingival preparation will be done to achieve a feather-edge finish line.
  Prepared tooth should be free from any blood or saliva. Try-in will be done using the pink crowns, to check the occlusion and Passive fit of the crown.
  The zirconia crown will be luted with type I glass ionemer cement. Consistent firm finger pressure will be applied during cementation, Any excess cement will be removed, and proper occlusion will be verified
  Arms: zerconia crown
Other: stainless steel crown — An appropriately sized preformed stainless-steel crown will be selected. Tooth preparation will involve using a tapered bur to reduce the occlusal surface by 1 to 1.5 mm, with interproximal reduction made on the mesial and distal sides. The selected crown size will be checked, and a trial fit will be conducted prior to cementation. Crimping pliers will be used, and the crown will be cemented with Type 1 glass ionomer cement.
  Any excess cement will be removed, and proper occlusion will be verified
  Arms: stainless steel crown

SUMMARY:
• the goal of this clinical trial is To evaluate the clinical effectiveness of bioflex crowns and zirconia crowns compared to stainless steel crowns when

* restoring primary molars 45 participant their age range between 6 and 8 years participated in this study. The participants are divided into three groups representing group (A) for Bioflx crown (n=15), group (B) for Zirconia crown (n=15) and group ( C) for Stainless steel crown(n=15).

Clinical success will be assessed according to the Modified United States Public Health Service Evaluation (USPHS) criteria regarding: crown retention ,marginal integrity, surface roughness and color change.

Also the periodontal health will be evaluated using gingival index and plaque index according to Silness and Loe. Moreover parental and child satisfaction

* will be evaluated

ELIGIBILITY:
Inclusion Criteria:

* Children who are free from any systemic disease.
* Cooperative children (positive/ definitely positive) according to Frankl's behavior rating scale.
* Children with good to fair oral hygiene according to Loe and Silness plaque index.
* Primary molars with deep carious lesion, that are indicated for pulpotomy and crown.
* Primary molars having two-thirds of root structure left radiographically
* Parents' willingness to participate through informed written consent

Exclusion Criteria:

* Children with oral parafunctional habits.
* Primary molars with bifurcation involvement
* Presence of abscess or fistula related to the selected tooth
* Primary molars with insufficient crown structure

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-11-10 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
gingival health | follow up at 3,6 and 9 months
  Evaluated using the gingival index according to Löe and Silness (1967), with scores of 0 (no inflammation), 1 (mild inflammation), 2 (moderate inflammation), and 3 (severe inflammation).

SECONDARY OUTCOMES:
plaque accumulation | 3,6 and 9 months
  Measured using the Löe and Silness index, was scored from 0 to 3 (0 = no plaque, 1=Soft debris covering not more than one third of the tooth surface, 2=Soft debris covering more than one third, but not more than two thirds, 3 =Soft debris covering more than two thirds of the tooth surface.
crown retention | 3,6 and 9 months
  Assessed using the USPHS criteria, where "Alpha" = the crown is intact, "Bravo" = Crown is chipped (small but noticible loss of material)but not enough to expose the underlyingdentin/base, and "Charlie" = sufficient loss of crown substance to expose the underlying dentin/base or complete loss of the crown
marginal integrity | 3,6 and 9 months
  Assessed using the USPHS criteria, where "Alpha" indicates that the Crown is completely adapted to the tooth. No visible gap. No explorer catch at the margins, "Bravo" indicates Explorer catch, There is no visible evidence of a gap into which the explorer could penetrate, "Charlie" indicates Explorer penetrates into a deep gap that exposes dentin
color change | 3,6 and 9 months
  Assessed using the USPHS criteria where alpha =no change in color and bravo= There is change in color when compared to the baseline
surface roughness | 3,6 and 9 months
  Assessed using the USPHS criteria Alpha= crown surface is smooth, Bravo= crown surface is slightly rough or has scratches, Charlie= Surface is deeply rough, with irregular scratches
parental satisfaction | 3,6 and 9 months
  The questionnaire for assessing parental satisfaction includes four main categories for rating the following parameters whether the child's oral health, appearance and masticatory function were improved after placement of the crowns. Criteria evaluated in the survey will include also the parent's perception of the color and retention of each crown.
  Responses will be recorded on a five-point Likert scale, ranging from 1 (not at all satisfied) to 5 (very satisfied).
child post-operative discomfort | immediately post-operative and 48 hours post-operative
  Post-operative pain will be assessed using the face pain scale modified from the Maunuksela et al scale(1987)Immediately after the dental procedure . It consists of three schematic faces with different facial expressions for happy face (1) , indifferent face (2) and sad crying face (3) representing:
  1. Satisfaction,
  2. Indifference ,
  3. Dissatisfaction .The same examiner will contact each parent or guardian after 48 hours to gather information about any complaints regarding sensitivity \ pain reported by the child.

CONTACTS AND LOCATIONS:
Locations (1):
- outpatient clinic of pediatric dentistry -faculty of dentistry- Alexandria university, Alexandria, Azarita, Egypt

IPD SHARING:
Plan to Share IPD: No
patient privacy

REFERENCES:
- [Background] Taran PK, Kaya MS. A Comparison of Periodontal Health in Primary Molars Restored with Prefabricated Stainless Steel and Zirconia Crowns. Pediatr Dent. 2018 Sep 15;40(5):334-339. PMID 30355428
- [Background] Clark L, Wells MH, Harris EF, Lou J. Comparison of Amount of Primary Tooth Reduction Required for Anterior and Posterior Zirconia and Stainless Steel Crowns. Pediatr Dent. 2016 Jan-Feb;38(1):42-6. PMID 26892214
- [Background] Salman N, Khattab N, Gomaa Y, Elheeny A. Parental satisfaction regarding two types of commercial crowns for restoring pulpotomized primary molars. Egypt Dent J . 2021;67:2915-21.
- [Background] Sai Sarath K, Murali G, Elangovan A, Kalaivanan D. Case series on personalized pediatric posterior Zirconia crowns: Case report. Int J Pedod Rehabil . 2022;7:46-50.
- [Background] Mittal GK, Verma A, Pahuja H, Agarwal S, Tomar H. Esthetic crowns in pediatric dentistry: A review. Int J Contemporary Medical Res. 2016;3:1280-2.
- [Background] Holsinger DM, Wells MH, Scarbecz M, Donaldson M. Clinical Evaluation and Parental Satisfaction with Pediatric Zirconia Anterior Crowns. Pediatr Dent. 2016;38(3):192-7. PMID 27306242